CLINICAL TRIAL: NCT03874156
Title: MUscle Side-Effects of Atorvastatin in Coronary Patients (MUSE) -a Randomized Controlled Trial
Brief Title: MUscle Side-Effects of Atorvastatin in Coronary Patients
Acronym: MUSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: The Hospital of Vestfold (Other); Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: REK 2018/2302
Record Dates: First submitted 2019-03-05; First posted 2019-03-14 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Statin Adverse Reaction
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized double-blinded placebo controlled cross-over phase 4 study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Atorvastatin 40 mg once daily
  Interventions: Drug: Atorvastatin 40mg
- Placebo group (Placebo Comparator): Matched placebo tablet once daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40mg — Oral tablet fabricated and labelled at Krageroe Tablettproduksjon AS
  Arms: Intervention group
Drug: Placebo Oral Tablet — Oral tablet fabricated and labelled at KrageroeTablettproduksjon AS
  Arms: Placebo group

SUMMARY:
The study aims to estimate the effect of atorvastatin on muscular symptom intensity in coronary patients with subjective statin-associated muscle symptoms (SAMS) and to determine the association with blood levels of atorvastatin and its metabolites, to obtain an objective marker for true SAMS. A randomized study will include 80 coronary patients with SAMS during ongoing atorvastatin therapy or previous muscle symptoms that led to discontinuation of atorvastatin. Patients will be randomized to 7-weeks treatment with atorvastatin 40 mg/day in the first period and matched placebo in the second 7-weeks period, or placebo in the first period and atorvastatin in the second period. A control group (n=40) without muscle symptoms will have 7 weeks open treatment with atorvastatin 40 mg/day. Blood samples will be collected at baseline and after each treatment period, and muscular symptom intensities will be rated by the patients weekly. The primary outcome is the difference in aggregated mean Visual Analogue Scale (VAS) scores between the last three weeks of atorvastatin treatment and of placebo treatment. The main purpose is to develop an objective marker for true SAMS, by comparing SAMS associated with blinded atorvastatin treatment with blood concentrations of atorvastatin and its metabolites. Diagnostic and discrimination performance will be determined. The study provides new clinical knowledge on SAMS in coronary patients and may contribute to more personalized statin treatment and monitoring, fewer side-effects and consequently improved adherence and lipid management in future practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* First or recurrent diagnosis (myocardial infarction) or treatments (Percutaneous Coronary Intervention [PCI] or Coronary Artery Bypass Graft operation [CABG]) for a coronary heart disease (CHD) event at least 6 months prior to study start and prescribed atorvastatin (irrespective of dose)
* Reporting muscle complaints (i.e. pain, weakness, tenderness, stiffness or cramp) that they attribute to atorvastatin therapy or atorvastatin discontinuation due to muscle complains
* Signed informed consent and expected cooperation of the patient according to International Council for Harmonisation/Good Clinical Practice and national/local regulations

Exclusion Criteria:

* First or recurrent diagnosis (myocardial infarction) or treatments (PCI or CABG) for a CHD event the a) past 12 months prior to study start in high risk patients (i.e. at least one of following comorbid conditions: systolic heart failure, >1 previous myocardial infarction, kidney failure, diabetes, and smokers) and b) the past 6 months prior to study start in low risk patients without any of the co-morbid conditions mentioned above and in patients who are not taking a statin at all

  . Patients with symptomatic peripheral artery disease and patients with familial hypercholesterolemia
* Patient has any contraindications for atorvastatin listed in the Summary of Product Characteristics (i.e. known hypersensitivity to the ingredients, acute liver failure/ Alanine Aminotransferase > 3 times upper limit of the normal range in blood at study start, pregnancy and breastfeeding)
* History of previous rhabdomyolysis, myopathy or liver failure due to statin treatment with Creatine Kinase > 10 times upper limit of the normal range or Alanine Aminotransferase > 3 times upper limit of the normal range.
* Any condition (e.g. psychiatric illness, dementia) or situation, that in the investigator's opinion could put the subject at significant risk, confound the study results, interfere significantly with the subject participation in the study, or rendering informed consent unfeasible
* Short life expectancy (<12 months) due to other medical conditions
* Not being able to understand Norwegian.
* Women of childbearing potential defined as all premenopausal female.
* Participation in another randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Individual mean difference in muscular symptom intensity measured with a 0 (no symptoms) to 10 (worst imaginable symptoms) Visual Analogue Scale (VAS) score between treatment periods with statin and placebo | 16 weeks following randomization
  Individual mean difference in muscular symptom (i.e. pain, aching, tenderness, stiffness, cramp and/or weakness) intensity between treatment periods with statin and placebo, reported by the patients over the last three weeks (i.e. week 4-7) measured with a 0 (no symptoms) to 10 (worst imaginable symptoms) Visual Analogue Scale (VAS) score with aggregated data from each subscale

SECONDARY OUTCOMES:
The proportion of patients who report muscle symptoms on atorvastatin treatment and not on placebo (dichotomous Statin Associated Muscle Symptom classification) | 16 weeks following randomization
The correlation between individual muscular symptom intensity between treatment periods with statin and placebo over the last three weeks measured with 0 to 10 VAS score aggregated from each subscale, and levels of atorvastatin and metabolites | 16 weeks following randomization
Sensitivity, specificity, and area under the curve of blood concentrations of parent drug and the active metabolites of atorvastatin for the classification of true Statin Associated Muscle Symptoms (SAMS) | 16 weeks following randomization
Individual mean difference in likelihood of statin discontinuation between treatment periods with statin and placebo over the last three weeks (i.e. week 4-7) measured with 0 to 10 VAS score with aggregated data from each subscale. | 16 weeks following randomization
Statin adherence measured weekly with self-reported questionnaire methods during the study periods | 16 weeks following randomization
  Statin adherence measured with self-reported questionnaires (numeric scale: <4/7, 5/7, 6/7 or 7/7) weekly during the treatment periods. Low statin adherence will be defined by taking statins less than 42 of 49 days during the 7 weeks treatment period
Statin adherence measured with pill counts of returned packages | 16 weeks following randomization
  Statin adherence measured with pill counts of returned packages. Low statin adherence will be defined by a total of >=8 returned pills during the treatment periods
Statin adherence measured with direct liquid chromatography-tandem mass spectrometry methods | 16 weeks following randomization
  Statin adherence measured with direct liquid chromatography-tandem mass spectrometry methods. Low statin adherence defined by dose-normalized statin and metabolites concentrations < 0.10 (nmol/L)/mg
Levels of atorvastatin and its metabolites in blood plasma and white blood cells at study end | 16 weeks following randomization
Number of patients with new-onset coronary heart disease symptoms, intolerable muscle symptoms leading to discontinuation from the treatment arm, and elevated levels of creatine kinase (CK) and/or Alanine Aminotransferase (ALT) in blood | 16 weeks following randomization
  Safety endpoints: i.New-onset coronary heart disease symptoms. ii Intolerable muscle symptoms leading to discontinuation from the treatment arm.iii elevated levels of creatine kinase (CK) and/or Alanine Aminotransferase (ALT) in blood

CONTACTS AND LOCATIONS:
Overall Officials: john munkhaugen, MD, PhD, Principal Investigator — Vestre Viken Trust
Locations (2):
- Norway (2):
  - Vestre Viken Trust, Drammen Hospital, Drammen, Buskerud
  - Hospital of Vestfold Trust, Tønsberg, Vestfold

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available for other researchers
Time Frame: Data will be available within 5 years of study completion

REFERENCES:
- [Derived] Sverre E, Munkhaugen J, Kristiansen O, Weedon-Fekjaer H, Peersen K, Gjertsen E, Gullestad L, Bergan S, Husebye E, Vethe NT. Plasma concentration of atorvastatin metabolites correlates with low-density lipoprotein cholesterol reduction in patients with coronary heart disease. Pharmacol Res Perspect. 2023 Jun;11(3):e01089. doi: 10.1002/prp2.1089. PMID 37186070

DOCUMENTS (2):
  • Study Protocol (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03874156/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03874156/SAP_001.pdf